CLINICAL TRIAL: NCT00926770
Title: Measurement of Cerebral Oxygenation With Near Infrared Spectroscopy During Blood Sampling From a Peripheral Artery Catheter in Preterm Infants With Gestational Age <37+0
Brief Title: Cerebral Near Infrared Spectroscopy During Blood Sampling From a Peripheral Artery Catheter in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: University of Cologne, Angela Kribs
Other Study IDs: 06-131
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Cerebral Oxygenation; Cerebral Blood Flow; Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pretem infants (GG < 37+0)

SUMMARY:
Preterm infants often need peripheral artery catheters for invasive blood pressure recording and to facilitate blood sampling. Near infrared spectroscopy is a method to evaluate cerebral oxygenation and as well as cerebral blood flow. Sampling procedures with identical sampling volumes are performed at a short (40 seconds) and a long (70 seconds) time intervall while changes of cerebral oxygenation are measured. The investigators hypothesise that slower sampling decrease changes in cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant (Gestational Age <37+0)
* Peripheral arterial catheter (ulnary or radial artery)

Exclusion Criteria:

* Complex organ malformation

Ages: 1 Minute to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants (Gestational Age <37+0)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-11

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cologne, NICU, Cologne, North Rhine-Westphalia, Germany